CLINICAL TRIAL: NCT01928940
Title: A Japanese Open-label Phase I/II Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of GSK2118436 and GSK1120212 Combination Therapy in Subjects With BRAF V600E/K Mutation Positive Advanced Solid Tumors (Phase I Part) and BRAF V600E/K Mutation Positive Cutaneous Melanoma (Phase II Part).
Brief Title: Japan PhI/II of GSK2118436 and GSK1120212 Combination in Subjects With BRAF V600E/K Mutation Positive Advanced Solid Tumors (Phase I Part) or Cutaneous Melanoma (Phase II Part)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116885
Record Dates: First submitted 2013-07-03; First posted 2013-08-27 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Solid Tumours
Keywords: Advanced solid tumors; BRAF; Melanoma
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dabrafenib + trametinib (Experimental): Combination therapy of dabrafenib and trametinib
  Interventions: Drug: dabrafenib; Drug: trametinib

INTERVENTIONS:
Drug: dabrafenib — 150 mg twice daily
Drug: trametinib — 2 mg once daily

SUMMARY:
This is a Japanese Phase I/II, open-label, non-controlled study to evaluate the safety, tolerability, pharmacokinetic profile, and efficacy of the combination of GSK2118436 and GSK1120212 in subjects with BRAF V600E/K mutation positive advanced solid tumors (Phase I part) and BRAF V600E/K mutation positive cutaneous melanoma (Phase II part).

DETAILED DESCRIPTION:
This is a Japanese Phase I/II, open-label, non-controlled study to evaluate the safety, tolerability, pharmacokinetic profile, and efficacy of the combination of GSK2118436 and GSK1120212 in subjects with BRAF V600E/K mutation positive advanced solid tumors (Phase I part) and BRAF V600E/K mutation positive cutaneous melanoma (Phase II part). Phase I part is designed to primarily assess the safety and tolerability of GSK2118436 and GSK1120212 combination therapy in subjects with BRAF V600E/K mutation positive advanced solid tumors. Six evaluable subjects will be enrolled into Phase I part and receive the combination therapy of GSK2118436 (150 mg, twice daily) and GSK1120212 (2 mg, once daily). A decision for starting Phase II part will be made by careful review based on available safety, tolerability and pharmacokinetic data in Phase I part. Phase II part is designed to primarily evaluate ORR of the combination as first-line therapy in subjects with unresectable (Stage IIIC) or metastatic (Stage IV) BRAF V600E/K mutation positive cutaneous melanoma. Subjects who have had prior systemic anti-cancer treatment in the advanced or metastatic setting will not be eligible for Phase II part although prior systemic treatment in the adjuvant setting will be allowed. Six evaluable subjects will be enrolled in Phase II part.

ELIGIBILITY:
Inclusion Criteria:

* Capable of given written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Male or female age 20 years or greater; able to swallow and retain oral medication.
* BRAF mutation positive advanced solid tumor ( Phase I part). BRAF mutation positive melanoma (Phase II part).
* Measurable disease according to RECIST version 1.1.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Agree to contraception requirements.
* Adequate organ system function.

Exclusion Criteria:

* Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy).
* Phase II part ONLY: Prior systemic anti-cancer treatment (chemotherapy, immunotherapy, biologic therapy, vaccine therapy, or investigational treatment) for Stage IIIC (unresectable) or Stage IV (metastatic) melanoma. Prior systemic treatment in the adjuvant setting is allowed.
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 28 days prior to the study treatment (6 weeks for prior nitrosourea or mitomycin C), or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to the study treatment. Limited radiotherapy within the last 2 weeks. (Note: Ipilimumab treatment must end at least 8 weeks prior to the study treatment.)
* Taken an investigational drug within 28 days or 5 half-lives (minimum 14 days), whichever is shorter, prior to the study treatment.
* Current use of a prohibited medication or requires any of these medications during treatment with the study drugs.
* A history of another malignancy. Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
* Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures (e.g., uncontrolled diabetes).
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs.
* History of pneumonitis or interstitial lung disease.
* Known HIV infection.
* Certain cardiac abnormality
* A history or current evidence/risk of retinal vein occlusion or central serous retinopathy.
* Pregnant or lactating female.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08-15; Primary Completion 2014-09-18 (Actual); Study Completion 2016-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of 2 parts: Phase I part included Japanese participants (par.) with BRAF V600E/K mutation-positive advanced solid tumors and the Phase II part included Japanese par. with BRAF V600E/K mutation-positive cutaneous melanoma.
Groups:
- Phase I: GSK2118436 150 mg + GSK1120212 2 mg: In the Phase I part, participants with BRAF V600E/K mutation-positive advanced solid tumors received the combination therapy of GSK2118436 150 milligrams (mg) (a combination of 75 mg capsules) orally twice daily (BID) and GSK1120212 2 mg tablet orally once daily (QD) until disease progression, death or an unacceptable adverse event. GSK2118436 and GSK1120212 were administered in the morning at approximately the same time. The second dose of GSK2118436 was taken in the evening approximately 12 hours (hr) after the morning dose. The second dose of GSK2118436 was not administered on Day 1 for the 24 hr serial pharmacokinetic (PK) blood sampling. Study drugs were taken with approximately 200 milliliters (mL) of water under fasting conditions, either 1 hr before or 2 hr after a meal.
- Phase II: GSK2118436 150 mg + GSK1120212 2 mg: In the Phase II part, participants with BRAF V600E/K mutation-positive cutaneous melanoma received the combination therapy of GSK2118436 150 mg (a combination of 75 mg capsules) orally BID and GSK1120212 2 mg tablet orally QD until disease progression, death or an unacceptable adverse event. GSK2118436 and GSK1120212 were administered in the morning at approximately the same time. The second dose of GSK2118436 was taken in the evening approximately 12 hr after the morning dose. Study drugs were taken with approximately 200 mL of water under fasting conditions, either 1 hr before or 2 hr after a meal.
Period: Overall Study
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg | Phase II: GSK2118436 150 mg + GSK1120212 2 mg | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (19.83) | 59.0 (10.99) | 55.6 (15.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 1 | 4 | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants With Any Adverse Event (AE) and Any Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence (MO) in a part. temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. SAE is defined as any untoward MO that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, a congenital anomaly/birth defect and protocol-specific SAEs:ALT>=3xupper limit of normal(ULN) and bilirubin>=2xULN(>35% direct) (or ALT>=3xULN, international normalized ratio>1.5), any new primary cancers, treatment emergent malignancies except basal cell carcinoma, symptomatic or asymptomatic LVEF decrease, retinal pigment epithelial detachment or retinal vein occlusion, pyrexia with hypotension,or dehydration or renal insufficiency,or severe (>=G3) rigor/chills.
Time Frame: From the start of study treatment until 30 days after study treatment discontinuation (average of 1.38 year)
Population: All Treated Subject (ATS) Population: all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Any AEs | 6
  Any SAEs | 1

2. Primary Outcome: Phase I: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: A DLT was defined as an event occurred during the first 21 days after the first dose of study drugs and met any of the following criteria, according to National Cancer Institutes (NCI) common terminology criteria for AE (CTCAE) grade (G) version 4.0: G4 hematological toxicity; G3 or G4 non-hematologic toxicity (including rash, nausea, vomiting and diarrhea only if uncontrolled with supportive therapy); rash >=G3 that required dose reduction despite supportive care; a G2 or greater non-hematological toxicity that in the judgment of the investigator and medical monitor; dose interruption of greater than 14 consecutive days due to unresolved toxicity; any new G2 or greater valvular heart disease and significant alteration in cardiac valve morphology from Baseline.
Time Frame: From the start of study treatment until 21 days
Population: DLT assessment Population: all participants for whom DLT assessment was appropriately conducted
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 5
Participants | 0

3. Primary Outcome: Phase I: Number of Participants With the Indicated Worst-case Change From Baseline (BL) in the Indicated Clinical Chemistry Parameters (CCPs)
Description: CCPs were graded according to NCI CTCAE grade version 4.0 as: G1, Mild; G2, Moderate; G3, Severe; G4, Life-threatening or disabling; G5, Death. Data are presented for only those parameters (para) for which an increase to G3 or G4 from BL G occurred. CCPs that were not G according to NCI CTCAE criteria, were categorized as High and Low with respect to the normal range. Data are presented only for those para for which the category decreased to Low or increased to High relative to the BL category. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments. CCPs included: albumin, alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, calcium, creatinine, glucose, potassium, magnesium, sodium, inorganic phosphorus, chloride, lactate dehydrogenase (LDH), total protein, urea/blood urea nitrogen (BUN) and uric acid.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 year)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Alkaline Phosphatase, G3 | 1
  ALT, G3 | 1
  Inorganic Phosphorous, G4 | 1
  Chloride, Low | 2
  LDH, Low | 1
  LDH, High | 3
  Total Protein, Low | 2
  Urea/BUN, Low | 1
  Urea/BUN, High | 2
  Uric acid, Low | 1
  Uric acid, High | 1

4. Primary Outcome: Phase I: Number of Participants With the Indicated Worst-case Change From Baseline in the Indicated Hematology Parameters
Description: Hematology parameters were summarized according to NCI CTCAE G, version 4.0 as: G1, Mild; G2, Moderate; G3, Severe; G4, Life-threatening or disabling; G5, Death. Data are presented for only those parameters for which an increase to G3 or G4 from Baseline G occurred. For hematology parameters that were not graded according to NCI CTCAE criteria, were categorized as High and Low with respect to the normal range. Data are presented only for those parameters for which the category decreased to Low or increased to High relative to the Baseline category. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments. Hematology parameters included: hemoglobin, lymphocytes, total neutrophils, platelet count, white blood cell (WBC) counts, basophils, eosinophils, hematocrit, mean corpuscular hemoglobin concentration (MCHC), mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), monocytes and red blood cell (RBC) count.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 year)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Lymphocytes, G3 | 1
  Total Neutrophils, G3 | 1
  Basophils, High | 1
  Eosinophils, High | 1
  Hematocrit, Low | 3
  MCHC, Low | 1
  MCH, Low | 2
  MCV, Low | 1
  Monocytes, Low | 2
  Monocytes, High | 3
  RBC count, Low | 4

5. Primary Outcome: Phase I: Number of Participants With the Indicated Urinalysis Parameters
Description: Urine samples were collected for urine dipstick analysis at Baseline and at the post-treatment Visit. The number of participants with negative (absence) and positive (presence: trace, 1+, 2+, 3+, 4+ or 5+) results for urine occult blood (UOB), urine glucose (UGLU), urine ketones (UKET), urine protein (UP) and urine urobilinogen (UUBIL) were summarized. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 year)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  UOB, Baseline, Negative | 6
  UOB, Baseline, Positive | 0
  UOB, Post-Treatment, Negative | 2
  UOB, Post-Treatment, Positive | 1
  UGLU, Baseline, Negative | 6
  UGLU, Baseline, Positive | 0
  UGLU, Post-Treatment, Negative | 3
  UGLU, Post-Treatment, Positive | 0
  UKET, Baseline, Negative | 6
  UKET, Baseline, Positive | 0
  UKET, Post-Treatment, Negative | 3
  UKET, Post-Treatment, Positive | 0
  UP, Baseline, Negative | 5
  UP, Baseline, Positive | 1
  UP, Post-Treatment, Negative | 2
  UP, Post-Treatment, Positive | 0
  UUBIL, Baseline, Negative | 0
  UUBIL, Baseline, Positive | 6
  UUBIL, Post-Treatment, Negative | 0
  UUBIL, Post-Treatment, Positive | 3

6. Primary Outcome: Phase I: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance (Pef) Status
Description: The ECOG pef status 5-point scale is used to assess how a participant's disease is progressing, to assess how the disease affects the daily living abilities of the par. and to determine appropriate treatment and prognosis: G0, fully active, able to carry on all pre-disease pef without restriction. G1, restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, example, light house work, office work. G2, ambulatory and capable of all selfcare, but unable to carry out any work activities; up and about >50 percent (%) of waking hrs. G3, capable of only limited selfcare; confined to bed or chair >50% of waking hrs. G4, completely disabled; cannot carry on any selfcare; totally confined to bed or chair. G5, dead. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments. Number of par. who improved, had no change, or deteriorated in pef status from BL is summarized.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 year)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Improved | 1
  No change | 4
  Deteriorated | 1

7. Primary Outcome: Phase I: Number of Participants With Worst-case On-therapy Increase From Baseline in Systolic and Diastolic Blood Pressure to Grade 2 or Grade 3
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) values were graded using (NCI CTCAE version 4.0). SBP was categorized as: G1 (Increase to >=120 to 140 millimeters of mercury [mmHg]), G2 (Increase to >=140 to <160 mmHg), and G3 (Increase to >=160 mmHg). DBP was categorized as: G1 (Increase to >=80 to <90 mmHg), G2 (Increase to >=90 to <100 mmHg), and G3 (Increase to >=100 mmHg). The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments. An increase is defined as an increase in the CTCAE grade relative to the Baseline grade. Participants with missing Baseline values were assumed to have a Baseline value of G0.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 year)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  SBP, Increase to Grade 2 | 3
  SBP, Increase to Grade 3 | 0
  DBP, Increase to Grade 2 | 2
  DBP, Increase to Grade 3 | 1

8. Primary Outcome: Phase I: Number of Participants With Worst-case On-therapy Change From Baseline in Heart Rate
Description: Change from Baseline in heart rate is categorized as decrease to <60 beats per minute (bpm), change to normal or no change, and increase to >100 bpm relative to the Baseline value. Participants with a missing Baseline value are assumed to have a normal Baseline value. Participants were counted twice if the participant's heart rate value decreased to <60 bpm and increased to >100 bpm post-Baseline. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 year)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Decrease to <60 bpm | 1
  Change to normal or no change | 3
  Increase to >100 bpm | 3

9. Primary Outcome: Phase I: Number of Participants With Worst-case On-therapy Change From Baseline in Temperature
Description: Change from Baseline in temperature is categorized as a decrease to <=35 degrees celsius (C), change to normal or no change as 35-38 degrees C, and increase to >=38 degrees C relative to the Baseline value. Participants with a missing Baseline value are assumed to have a normal Baseline value. Participants were counted twice if the participant temperature value decreased to <=35 degrees C and increased to >=38 degrees C post-Baseline. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Decrease to <=35 degrees C | 2
  Change to normal or no change | 2
  Increase to >=38 degrees C | 3

10. Primary Outcome: Phase I: Change From Baseline in Oxygen Saturation (SpO2) Measured Via Pulse Oxymetry at the Indicated Time Points
Description: Oxygen saturation measures the capacity of blood to transport oxygen to other parts of the body. Oxygen binds to hemoglobin in red blood cells when moving through the lungs. A pulse oximeter uses two frequencies of light (red and infrared) to determine the percentage of hemoglobin in the blood that is saturated with oxygen,that is called as blood oxygen saturation or SpO2. Change from Baseline was calculated as the individual post-Baseline value (Days 8,15; Weeks 3 to 136 and post-treatment Visit) minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 year)
Population: ATS Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Percentage of oxygen in blood
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Percentage of oxygen in blood
  Day 8, n=6 | 1.0 (0.89)
  Day 15, n=6 | 0.8 (0.75)
  Week 3, n=6 | 0.2 (0.75)
  Week 8, n=6 | 0.7 (1.21)
  Week 12, n=5 | 1.4 (1.67)
  Week 16, n=6 | 1.2 (2.14)
  Week 20, n=5 | 0.4 (1.14)
  Week 24, n=5 | 0.8 (1.92)
  Week 28, n=5 | 0.8 (1.92)
  Week 32, n=5 | 0.6 (1.14)
  Week 36, n=5 | 0.8 (1.30)
  Week 40, n=4 | 0.5 (1.00)
  Week 44, n=4 | 0.5 (2.38)
  Week 48, n=4 | 0.5 (2.08)
  Week 52, n=2 | -0.5 (2.12)
  Week 56, n=2 | 0.0 (0.00)
  Week 60, n=2 | -0.5 (0.71)
  Week 64, n=2 | 0.0 (0.00)
  Week 68, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 72, n=1 | 1.0 (NA) — There were too few participants to provide a dispersion value.
  Week 76, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 80, n=1 | 1.0 (NA) — There were too few participants to provide a dispersion value.
  Week 84, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 88, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 92, n=1 | -2.0 (NA) — There were too few participants to provide a dispersion value.
  Week 96, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 100, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 104, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 108, n=1 | -1.0 (NA) — There were too few participants to provide a dispersion value.
  Week 112, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 116, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 120, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 124, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 128, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 132, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Week 136, n=1 | 0.0 (NA) — There were too few participants to provide a dispersion value.
  Post-Treatment, n=4 | 0.8 (0.96)

11. Primary Outcome: Phase I: Change From Baseline in Weight at the Indicated Time Points
Description: Mean change in body weight from Baseline was determined. Change from Baseline was calculated as the individual post-Baseline value (Weeks 3 to 136 and post-treatment Visit) minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: From Baseline until the post-treatment Visit ( average of 1.38 year)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Kilogram (Kg)
  Week 3, n=6 | -4.87 (6.046)
  Week 8, n=6 | -4.43 (6.274)
  Week 12, n=6 | -4.13 (6.436)
  Week 16, n=6 | -4.00 (6.801)
  Week 20, n=5 | -0.62 (2.295)
  Week 24, n=5 | -0.70 (1.402)
  Week 28, n=5 | -0.36 (1.850)
  Week 32, n=5 | -0.38 (1.809)
  Week 36, n=5 | -0.78 (1.821)
  Week 40, n=4 | -1.43 (1.305)
  Week 44, n=4 | -0.68 (1.759)
  Week 48, n=4 | -1.03 (2.081)
  Week 52, n=2 | 0.15 (2.475)
  Week 56, n=2 | -0.30 (1.556)
  Week 60, n=2 | -0.35 (2.475)
  Week 64, n=2 | -0.05 (2.475)
  Week 68, n=1 | -2.60 (NA) — There were too few participants to provide a dispersion value.
  Week 72, n=1 | -2.10 (NA) — There were too few participants to provide a dispersion value.
  Week 76, n=1 | -1.20 (NA) — There were too few participants to provide a dispersion value.
  Week 80, n=1 | -0.70 (NA) — There were too few participants to provide a dispersion value.
  Week 84, n=1 | -0.70 (NA) — There were too few participants to provide a dispersion value.
  Week 88, n=1 | -1.20 (NA) — There were too few participants to provide a dispersion value.
  Week 92, n=1 | -0.80 (NA) — There were too few participants to provide a dispersion value.
  Week 96, n=1 | -0.80 (NA) — There were too few participants to provide a dispersion value.
  Week 100, n=1 | -0.80 (NA) — There were too few participants to provide a dispersion value.
  Week 104, n=1 | -0.50 (NA) — There were too few participants to provide a dispersion value.
  Week 108, n=1 | -1.00 (NA) — There were too few participants to provide a dispersion value.
  Week 112, n=1 | -1.00 (NA) — There were too few participants to provide a dispersion value.
  Week 116, n=1 | -0.50 (NA) — There were too few participants to provide a dispersion value.
  Week 120, n=1 | -0.60 (NA) — There were too few participants to provide a dispersion value.
  Week 124, n=1 | -0.70 (NA) — There were too few participants to provide a dispersion value.
  Week 128, n=1 | -0.60 (NA) — There were too few participants to provide a dispersion value.
  Week 132, n=1 | -0.80 (NA) — There were too few participants to provide a dispersion value.
  Week 136, n=1 | -0.50 (NA) — There were too few participants to provide a dispersion value.
  Post-Treatment, n=4 | -0.05 (1.457)

12. Primary Outcome: Phase I: Number of Participants With the Indicated Electrocardiogram (ECG) Findings at the Indicated Time Points
Description: Single twelve (12)-lead ECGs were perfomred at Baseline, Weeks 3 to 132 and post-treatment Visit. ECG findings were categorized as: normal, abnormal - clinically significant (CS), or abnormal - not clinically significant (NCS), as determined by the investigator.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 year)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Baseline, Normal, n=6 | 4
  Baseline, Abnormal-NCS, n=6 | 2
  Baseline, Abnormal-CS, n=6 | 0
  Week 3, Normal, n=6 | 5
  Week 3, Abnormal-NCS, n=6 | 1
  Week 3, Abnormal-CS, n=6 | 0
  Week 12, Normal, n=6 | 5
  Week 12, Abnormal-NCS, n=6 | 1
  Week 12, Abnormal-CS, n=6 | 0
  Week 24, Normal, n=5 | 4
  Week 24, Abnormal-NCS, n=5 | 1
  Week 24, Abnormal-CS, n=5 | 0
  Week 36, Normal, n=5 | 4
  Week 36, Abnormal-NCS, n=5 | 1
  Week 36, Abnormal-CS, n=5 | 0
  Week 48, Normal, n=4 | 2
  Week 48, Abnormal-NCS, n=4 | 2
  Week 48, Abnormal-CS, n=4 | 0
  Week 60, Normal, n=2 | 2
  Week 60, Abnormal-NCS, n=2 | 0
  Week 60, Abnormal-CS, n=2 | 0
  Week 72, Normal, n=1 | 1
  Week 72, Abnormal-NCS, n=1 | 0
  Week 72, Abnormal-CS, n=1 | 0
  Week 84, Normal, n=1 | 1
  Week 84, Abnormal-NCS, n=1 | 0
  Week 84, Abnormal-CS, n=1 | 0
  Week 96, Normal, n=1 | 1
  Week 96, Abnormal-NCS, n=1 | 0
  Week 96, Abnormal-CS, n=1 | 0
  Week 108, Normal, n=1 | 1
  Week 108, Abnormal-NCS, n=1 | 0
  Week 108, Abnormal-CS, n=1 | 0
  Week 120, Normal, n=1 | 1
  Week 120, Abnormal-NCS, n=1 | 0
  Week 120, Abnormal-CS, n=1 | 0
  Week 132, Normal, n=1 | 1
  Week 132, Abnormal-NCS, n=1 | 0
  Week 132, Abnormal-CS, n=1 | 0
  Post-Treatment, Normal, n=3 | 3
  Post-Treatment, Abnormal-NCS, n=3 | 0
  Post-Treatment, Abnormal-CS, n=3 | 0

13. Primary Outcome: Phase I: Number of Participants With Worst-case On-therapy Change From Baseline in Left Ventricular Ejection Fraction (LVEF) as Assessed by Echocardiogram (ECHO)
Description: Absolute change from Baseline in LVEF were summarized at each scheduled assessment time and in the worst-case post Baseline. Only the post Baseline assessments that used the same method (ECHO or Multi Gated Acquisition Scan [MUGA]) as the Baseline assessments were used to derive the change from Baseline. The change from Baseline was categorized as: any increase; no change; 0-<10 Decrease, 10-19 Decrease, >=20 Decrease, >=10 Decrease and >= lower limit of normal (LLN), >=10 Decrease and below LLN, >=20 Decrease and >=LLN and >=20 Decrease and below LLN. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Any Increase | 0
  No change | 0
  0-<10 Decrease | 5
  10-19 Decrease | 1
  >=20 Decrease | 0
  >=10 Decrease and >=LLN | 1
  >=10 Decrease and below LLN | 0
  >=20 Decrease and >=LLN | 0
  >=20 Decrease and below LLN | 0

14. Primary Outcome: Phase II: Number of Participant With Confirmed Overall Response
Description: Confirmed overall response (ORR) is defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. RECIST is a set of rules that define when tumors in cancer participants improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment. CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions after treatment from Baseline (before study drug administration). ORR was assessed by investigator and blinded independent central review (BICR).
Time Frame: Every 8 weeks from start of the treatment until disease progression, death, or withdrawal of consent (average of 1.38 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Investigator-Assessed | 5
  BICR-Assessed | 5
Statistical Analysis 1: Comparison: Phase II: GSK2118436 150 mg + GSK1120212 2 mg; Test type: Superiority or Other; p < 0.0001, Exact binomial test; Percentage = 83, 95% CI 2-sided [35.9 to 99.6] — For Investigator Assessed ORR
Statistical Analysis 2: Comparison: Phase II: GSK2118436 150 mg + GSK1120212 2 mg; Test type: Superiority or Other; p < 0.0001, Exact binomial test; Percentage = 83, 95% CI 2-sided [35.9 to 99.6] — BICR Assessed ORR

15. Secondary Outcome: Phase I: Area Under the Plasma Concentration Versus Time Curve (AUC) of GSK2118436 and Metabolites, and GSK1120212 After Single and Repeat Dose
Description: Blood samples were collected from each par. at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hr after administration of GSK2118436 + GSK1120212 on Day 1 (single dose) and at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hr post-dose on Day 21 (repeat dose) for PK analysis. GSK2118436 metabolites included GSK2285403, GSK2298683, and GSK2167542. AUC from time zero to last quantifiable concentration (concn) (AUC[0-t]) was determined using the linear trapezoidal rule for increasing concn and the logarithmic trapezoidal rule for decreasing. The AUC from time zero extrapolated to infinity (AUC[0-inf] was calculated, where data permit, as the sum of AUC(0-t) and Ct/z, where Ct is the observed plasma concn obtained from the log-linear regression analysis of the last quantifiable time-point and z is the terminal phase rate constant. Area under the concentration-time curve over 12 hr and 24 hr dosing interval is called AUC[0-12] and AUC[0-24]. AUC(0-inf) was calculated only at Day 1.
Time Frame: At pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hr after administration of GSK2118436 + GSK1120212 on Day 1 (single dose) and at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hr on Day 21 (repeat dose)
Population: PK Population: all par. included in the ATS population for whom a PK sample was obtained and analyzed. Only those par. available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nanogram (ng)/mL
Groups:
- Phase I: GSK2118436 150 mg + GSK1120212 2 mg: In the Phase I part, participants with BRAF V600E/K mutation-positive advanced solid tumors received the combination therapy of GSK2118436 150 mg (a combination of 75 mg capsules) orally BID and GSK1120212 2 mg tablet orally QD until disease progression, death or an unacceptable adverse event. GSK2118436 and GSK1120212 were administered in the morning at approximately the same time. The second dose of GSK2118436 was taken in the evening approximately 12 hr after the morning dose. The second dose of GSK2118436 was not administered on Day 1 for the 24 hr serial PK blood sampling. Study drugs were taken with approximately 200 mL of water under fasting conditions, either 1 hr before or 2 hr after a meal.
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
hr*nanogram (ng)/mL
  GSK2118436, AUC[0-t], Day 1, n=6 | 12850.5346 (37.3)
  GSK2118436, AUC[0-t], Day 21, n=6 | 10075.3530 (32.4)
  GSK2118436, AUC[0-12], Day 1, n=6 | 11414.9211 (41.3)
  GSK2118436, AUC[0-12], Day 21, n=6 | 10138.0887 (33.1)
  GSK2118436, AUC[0-inf], Day 1, n=6 | 13485.6357 (36.9)
  GSK2285403, AUC[0-t], Day 1, n=6 | 10530.0297 (39.4)
  GSK2285403, AUC[0-t], Day 21, n=6 | 7199.9862 (29.9)
  GSK2285403, AUC[0-12], Day 1, n=6 | 7929.4506 (64.3)
  GSK2285403, AUC[0-12], Day 21, n=6 | 7273.0445 (30.6)
  GSK2285403, AUC[0-inf], Day 1, n=6 | 13903.4979 (67.9)
  GSK2298683, AUC[0-t], day 1, n=6 | 50834.2106 (106.0)
  GSK2298683, AUC[0-t], Day 21, n=6 | 108578.495 (36.1)
  GSK2298683, AUC[0-12], Day 1, n=6 | 18963.4767 (255.7)
  GSK2298683, AUC[0-12], Day 21, n=6 | 113205.044 (36.8)
  GSK2298683, AUC[0-inf], Day 1, n=5 | 125748.810 (41.8)
  GSK2167542, AUC[0-t], Day 1, n=6 | 571.5619 (170.4)
  GSK2167542, AUC[0-t], Day 21, n=6 | 2503.0667 (92.7)
  GSK2167542, AUC[0-12], Day 1, n=6 | 116.1860 (269.6)
  GSK2167542, AUC[0-12], Day 21, n=4 | 2755.2522 (122.0)
  GSK2167542, AUC[0-inf], Day 1, n=1 | 4628.4351 (NA) — There were too few participants to provide a dispersion value
  GSK1120212, AUC[0-t], Day 1, n=6 | 69.3090 (50.2)
  GSK1120212, AUC[0-t], Day 21, n=6 | 261.2787 (20.9)
  GSK1120212, AUC[0-24], Day 1, n=5 | 82.5215 (23.1)
  GSK1120212, AUC[0-24], Day 21, n=6 | 447.9452 (25.5)
  GSK1120212, AUC[0-inf], Day 1, n=5 | 375.5275 (23.1)

16. Secondary Outcome: Phase I: Maximum Plasma Concentration (Cmax) of GSK2118436 and Metabolites, and GSK1120212 After a Single and Repeat Dose
Description: Blood samples were collected from each participant at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hr after administration of GSK2118436 + GSK1120212 on Day 1 (single dose) and at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hr post-dose on Day 21 (repeat dose) for PK analysis. GSK2118436 metabolites included GSK2285403, GSK2298683 and GSK2167542. Cmax was determined from the raw concentration-time data.
Time Frame: as for outcome 15
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
ng/mL
  GSK2118436, Day 1 | 2497.383 (69.7)
  GSK2118436, Day 21 | 3431.280 (12.0)
  GSK2285403, Day 1 | 1336.296 (70.1)
  GSK2285403, Day 21 | 1995.847 (14.8)
  GSK2298683, Day 1 | 3689.039 (75.5)
  GSK2298683, Day 21 | 12303.403 (32.5)
  GSK2167542, Day 1 | 50.405 (149.7)
  GSK2167542, Day 21 | 323.863 (82.4)
  GSK1120212, Day 1 | 7.824 (112.1)
  GSK1120212, Day 21 | 32.522 (20.2)

17. Secondary Outcome: Phase I: Plasma Trough Concentration (Ctau) of GSK2118436 and Metabolites, and GSK1120212 After a Single and Repeat Dose
Description: Trough concentration is the lowest level that a drug is present in the body. Pre-dose (trough) blood samples were collected on Day 8, Day 15, Weeks 3, 8, 16 and 24 for estimating plasma trough concentration. GSK2118436 metabolites included GSK2285403, GSK2298683, and GSK2167542. Ctau was determined from the raw concentration-time data.
Time Frame: At pre-dose on Day 8, Day 15, Weeks 3, 8, 16 and 24
Population: PK Population.Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
ng/mL
  GSK2118436, Day 8, n=6 | 118.36 (188.3)
  GSK2118436, Day 15, n=6 | 84.25 (136.2)
  GSK2118436, Week 3, n=6 | 78.14 (149.3)
  GSK2118436, Week 8, n=6 | 78.29 (591.4)
  GSK2118436, Week 16, n=6 | 105.05 (206.4)
  GSK2118436, Week 24, n=5 | 121.85 (183.9)
  GSK2285403, Day 8, n=6 | 149.61 (111.9)
  GSK2285403, Day 15, n=6 | 106.09 (72.8)
  GSK2285403, Week 3, n=6 | 93.87 (82.0)
  GSK2285403, Week 8, n=6 | 89.12 (239.4)
  GSK2285403, Week 16, n=6 | 100.10 (121.8)
  GSK2285403, Week 24, n=5 | 117.93 (121.4)
  GSK2298683, Day 8, n=6 | 6011.00 (39.8)
  GSK2298683, Day 15, n=6 | 5141.38 (39.5)
  GSK2298683, Week 3, n=6 | 6210.90 (51.8)
  GSK2298683, Week 8, n=6 | 4408.24 (65.0)
  GSK2298683, Week 16, n=6 | 4022.93 (39.4)
  GSK2298683, Week 24, n=5 | 4294.86 (51.9)
  GSK2167542, Day 8, n=6 | 217.73 (46.7)
  GSK2167542, Day 15, n=6 | 161.11 (107.5)
  GSK2167542, Week 3, n=6 | 224.32 (83.6)
  GSK2167542, Week 8, n=6 | 220.93 (52.2)
  GSK2167542, Week 16, n=6 | 270.15 (107.5)
  GSK2167542, Week 24, n=5 | 227.75 (101.5)
  GSK1120212, Day 8, n=6 | 11.36 (43.0)
  GSK1120212, Day 15, n=6 | 12.47 (22.4)
  GSK1120212, Week 3, n=6 | 13.80 (25.6)
  GSK1120212, Week 8, n=6 | 14.52 (65.0)
  GSK1120212, Week 16, n=6 | 13.47 (39.4)
  GSK1120212, Week 24, n=5 | 13.72 (41.3)

18. Secondary Outcome: Phase I: Time of Occurrence of Cmax (Tmax) and Terminal Phase Half Life (t1/2) of GSK2118436 and Metabolites, and GSK1120212 After a Single and Repeat Dose
Description: Blood samples were collected from each participant at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hr after administration of GSK2118436 + GSK1120212 on Day 1 (single dose) and at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 12 hr post-dose on Day 21 (repeat dose) for PK analysis. GSK2118436 metabolites included GSK2285403, GSK2298683, and GSK2167542. Tmax is defined as the time of occurrence of Cmax. Tmax was determined directly from the raw concentration-time data. The apparent terminal elimination half-life (t1/2) obtained as the ratio of ln2/lamdaz, where lamdaz is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data. . T1/2 was calculated only at Day 1.
Time Frame: as for outcome 15
Population: PK Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles)
Measure: Median (Full Range); unit: hr
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
hr
  GSK2118436, t1/2, Day 1, n=6 | 4.5398 [2.776 to 9.645]
  GSK2118436, tmax, Day 1, n=6 | 2.425 [1.43 to 3.85]
  GSK2118436, tmax, Day 21, n=6 | 1.685 [0.97 to 1.97]
  GSK2285403, t1/2, Day 1, n=6 | 4.2086 [3.574 to 55.294]
  GSK2285403, tmax, Day 1, n=6 | 3.410 [2.93 to 11.93]
  GSK2285403, tmax, Day 21, n=6 | 1.950 [1.47 to 2.93]
  GSK2298683, t1/2, Day 1, n=5 | 15.5414 [11.652 to 21.159]
  GSK2298683, tmax, Day 1, n=6 | 9.840 [7.92 to 23.82]
  GSK2298683, tmax, Day 21, n=6 | 4.955 [2.75 to 5.98]
  GSK2167542, t1/2, Day 1, n=1 | 55.8643 [55.8643 to 55.8643]
  GSK2167542, tmax, Day 1, n=6 | 23.885 [11.65 to 24.28]
  GSK2167542, tmax, Day 21, n=6 | 4.505 [1.97 to 9.92]
  GSK1120212, t1/2, Day 1, n=5 | 89.5954 [39.029 to 126.331]
  GSK1120212, tmax, Day 1, n=6 | 0.965 [0.92 to 23.82]
  GSK1120212, tmax, Day 21, n=6 | 1.210 [0.92 to 5.93]

19. Secondary Outcome: Phase I: Number of Participants With Confirmed Overall Response Rate
Description: Confirmed ORR is defined as the percentage of participants with a confirmed CR or PR according to RECIST, version 1.1. RECIST is a set of rules that define when tumors in cancer participants improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment. CR is defined as the disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions after treatment from Baseline (before study drug administration). ORR was assessed by investigator and BICR.
Time Frame: as for outcome 14
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Investigator-Assessed | 5
  BICR-Assessed | 3
Statistical Analysis 1: Comparison: Phase I: GSK2118436 150 mg + GSK1120212 2 mg; Test type: Superiority or Other; p < 0.0001, Exact binomial test; Percentage = 83, 95% CI 2-sided [35.9 to 99.6] — For Investigator Assessed ORR
Statistical Analysis 2: Comparison: Phase I: GSK2118436 150 mg + GSK1120212 2 mg; Test type: Superiority or Other; p = 0.0158, Exact binomial test; Percentage = 50, 95% CI 2-sided [11.8 to 82.2] — BICR Assessed ORR

20. Secondary Outcome: Phase I: Number of Participants With Unconfirmed Overall Response Rate
Description: ORR is defined as the percentage of participants with an unconfirmed CR or PR according to RECIST version 1.1. RECIST is a set of rules that define when tumors in cancer participants improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment. CR is defined as disappearance of all target lesions. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions after treatment from Baseline (before study drug administration). Unconfirmed ORR was assessed by investigator and BICR.
Time Frame: as for outcome 14
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Investigator-Assessed | 5
  BICR-Assessed | 3
Statistical Analysis 1: Comparison: Phase I: GSK2118436 150 mg + GSK1120212 2 mg; Test type: Superiority or Other; p < 0.0001, Exact binomial test; Percentage = 83, 95% CI 2-sided [35.9 to 99.6] — For Investigator Assessed ORR
Statistical Analysis 2: Comparison: Phase I: GSK2118436 150 mg + GSK1120212 2 mg; Test type: Superiority or Other; p = 0.0158, Exact binomial test; Percentage = 50, 95% CI 2-sided [11.8 to 88.2] — BICR Assessed ORR

21. Secondary Outcome: Phase I: Progression Free Survival (PFS)
Description: PFS is defined as the time from the first dose of study treatment to the earliest date of disease progression or death due to any cause. The length of this interval is estimated as the date of death or disease progression minus the date of first dose plus one day. The date of documented disease progression is defined as the date of disease progression based on radiologic evidence. Participants with documented date of disease progresssion or death and who had not received subsequent anticancer treatment prior to the date of documented disease progression or death were included in the analysis of PFS. PFS was assessed by investigator and BICR. Please note the values of the Full Range (min, max) are described irregardless of censoring at data cut-off.
Time Frame: From start of the treatment until disease progression or death (average of 1.38 years)
Population: ATS Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ATS population.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Weeks
  Investigator-Assessed, n=6 | NA [16 to 65.1] — The median values were not planned to calculate in the study analysis plan because lack of events had been estimated at the time of this primary analysis of the ORR.
  BICR-Assessed, n=6 | NA [9 to 65.1] — The median values were not planned to calculate in the study analysis plan because lack of events had been estimated at the time of this primary analysis of the ORR.

22. Secondary Outcome: Phase I: Duration of Response
Description: Duration of response is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause among participants with confirmed CR or PR. The participant who showed a CR or PR was included in the analysis of duration of response. Duration of response was assessed by investigator and BICR. Please note the values of the Full Range (min, max) are described irregardless of censoring at data cut-off.
Time Frame: From start of the treatment until disease progression or death (average of 1.38 years)
Population: as for outcome 21
Measure: Median (Full Range); unit: Weeks
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Weeks
  Investigator-Assessed, n=5 | NA [17.4 to 57.1] — The median values were not planned to calculate in the study analysis plan because lack of events had been estimated at the time of this primary analysis of the ORR.
  BICR-Assessed, n=3 | NA [32.1 to 57.1] — The median values were not planned to calculate in the study analysis plan because lack of events had been estimated at the time of this primary analysis of the ORR.

23. Secondary Outcome: Phase II: Number of Participants With Unconfirmed Overall Response
Description: as for outcome 20
Time Frame: as for outcome 14
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Investigator-Assessed | 5
  BICR-Assessed | 5
Statistical Analysis 1: Comparison: Phase II: GSK2118436 150 mg + GSK1120212 2 mg; Test type: Superiority or Other; p < 0.0001, Exact binomial test; Percentage = 83, 95% CI 2-sided [35.9 to 99.6] — For Investigator Assessed ORR
Statistical Analysis 2: Comparison: Phase II: GSK2118436 150 mg + GSK1120212 2 mg; Test type: Superiority or Other; p < 0.0001, Exact binomial test; Percentage = 83, 95% CI 2-sided [35.9 to 99.6] — BICR Assessed ORR

24. Secondary Outcome: Phase II: Progression Free Survival (PFS)
Description: as for outcome 21
Time Frame: From start of the treatment until disease progression or death (average of 1.38 years)
Population: as for outcome 21
Measure: Median (Full Range); unit: Weeks
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Weeks
  Investigator-Assessed, n=6 | NA [19.0 to 128.4] — The median values were not planned to calculate in the study analysis plan because lack of events had been estimated at the time of this primary analysis of the ORR.
  BICR-Assessed, n=6 | NA [19.0 to 128.4] — The median values were not planned to calculate in the study analysis plan because lack of events had been estimated at the time of this primary analysis of the ORR.

25. Secondary Outcome: Phase II: Duration of Response
Description: as for outcome 22
Time Frame: From start of the treatment until disease progression or death (average of 1.38 years)
Population: as for outcome 21
Measure: Median (Full Range); unit: Weeks
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Weeks
  Investigator-Assessed, n=5 | NA [16 to 120.1] — There were too few participants to provide a median PFS
  BICR-Assessed, n=5 | NA [11.1 to 120.1] — There were too few participants to provide a median PFS

26. Secondary Outcome: Phase II: Number of Participants With Any Adverse Event and Any Serious Adverse Event
Description: An AE is defined as any untoward MO in a part. temporally associated with the use of a MP, whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. SAE is defined as any untoward MO that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, a congenital anomaly/birth defect and protocol-specific SAEs:ALT>=3xULN and bilirubin>=2xULN(>35% direct) (or ALT>=3xULN, international normalized ratio>1.5), any new primary cancers, treatment emergent malignancies except basal cell carcinoma, symptomatic or asymptomatic LVEF decrease, retinal pigment epithelial detachment or retinal vein occlusion, pyrexia with hypotension,or dehydration or renal insufficiency,or severe (>=G3) rigor/chills.
Time Frame: From the start of study treatment until 30 days after study treatment discontinuation (average of 1.38 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Any AE | 6
  Any SAE | 0

27. Secondary Outcome: Phase II: Number of Participants With the Indicated Worst-case Change From Baseline in the Indicated Clinical Chemistry Parameters
Description: CCPs were graded according to NCI CTCAE garde version 4.0 as: G1, Mild; G2, Moderate; G3, Severe; G4, Life-threatening or disabling; G5, Death. Data are presented for only those parameters for which an increase to G3 or G4 from Baseline grade occurred. CCPs that were not graded according to NCI CTCAE criteria, were categorized as High and Low with respect to the normal range. Data are presented only for those parameters for which the category decreased to Low or increased to High relative to the Baseline category. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments. CCPs included: albumin, alkaline phosphatase, ALT, AST, total bilirubin, calcium, creatinine, glucose, potassium, magnesium, sodium, inorganic phosphorus, chloride, LDH, total protein, urea/BUN and uric acid.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Inorganic Phosphorous, G3 | 2
  Chloride, High | 2
  LDH, High | 5
  Total Protein, Low | 2
  Urea/BUN, High | 1
  Uric acid, Low | 1

28. Secondary Outcome: Phase II: Number of Participants With the Indicated Worst-case Change From Baseline in the Indicated Hematology Parameters
Description: Hematology parameters were summarized according to NCI CTCAE G, version 4.0 as: G1, Mild; G2, Moderate; G3, Severe; G4, Life-threatening or disabling; G5, Death. Data are presented for only those parameters for which an increase to G3 or G4 from Baseline G occurred. For hematology parameters that were not graded according to NCI CTCAE criteria, were categorized as High and Low with respect to the normal range. Data are presented only for those parameters for which the category decreased to Low or increased to High relative to the Baseline category. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments. Hematology parameters included: hemoglobin, lymphocytes, total neutrophils, platelet count, WBC counts, basophils, eosinophils, hematocrit, MCHC, MCH, MCV, monocytes and RBC count.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Total Neutrophils, G3 | 1
  Eosinophils, High | 1
  Hematocrit, Low | 2
  MCHC, Low | 1
  MCH, Low | 1
  MCV, Low | 1
  MCV, High | 1
  Monocytes, Low | 3
  Monocytes, High | 4
  RBC count, Low | 1
  RBC count, High | 1

29. Secondary Outcome: Phase II: Number of Participants With the Indicated Urinalysis Results
Description: Urine samples were collected for urine dipstick analysis at Baseline and at the post-treatment Visit. The number of participants with negative (absence) and positive (presence: trace, 1+, 2+, 3+, 4+ or 5+) results for UOB, UGLU, UKET, UP and UUBIL were summarized. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  UOB, Baseline, Negative | 6
  UOB, Baseline, Positive | 0
  UOB, Post-Treatment, Negative | 3
  UOB, Post-Treatment, Positive | 0
  UGLU, Baseline, Negative | 6
  UGLU, Baseline, Positive | 0
  UGLU, Post-Treatment, Negative | 2
  UGLU, Post-Treatment, Positive | 1
  UKET, Baseline, Negative | 5
  UKET, Baseline, Positive | 1
  UKET, Post-Treatment, Negative | 2
  UKET, Post-Treatment, Positive | 1
  UP, Baseline, Negative | 6
  UP, Baseline, Positive | 0
  UP, Post-Treatment, Negative | 2
  UP, Post-Treatment, Positive | 1
  UUBIL, Baseline, Negative | 0
  UUBIL, Baseline, Positive | 6
  UUBIL, Post-Treatment, Negative | 0
  UUBIL, Post-Treatment, Positive | 3

30. Secondary Outcome: Phase II: Number of Participants With the Indicated Worst-case On-therapy Change From Baseline in ECOG Perormance Status
Description: The ECOG pef status 5-point scale is used to assess how a participant's disease is progressing, to assess how the disease affects the daily living abilities of the par. and to determine appropriate treatment and prognosis: G0, fully active, able to carry on all pre-disease pef without restriction. G1, restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, example, light house work, office work. G2, ambulatory and capable of all selfcare, but unable to carry out any work activities; up and about >50% of waking hrs. G3, capable of only limited selfcare; confined to bed or chair >50% of waking hrs. G4, completely disabled; cannot carry on any selfcare; totally confined to bed or chair. G5, dead. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments. Number of par. who improved, had no change, or deteriorated in pef status from BL is summarized.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Improved | 0
  No change | 4
  Deteriorated | 2

31. Secondary Outcome: Phase II: Number of Participants With Worst-case On-therapy Increase From Baseline in Systolic and Diastolic Blood Pressure to Grade 2 or Grade 3
Description: SBP and DBP values were graded using (NCI CTCAE version 4.0). SBP was categorized as: G1 (Increase to >=120 to 140 mmHg), G2 (Increase to >=140 to <160 mmHg), and G3 (Increase to >=160 mmHg). DBP was categorized as: G1 (Increase to >=80 to <90 mmHg), G2 (Increase to >=90 to <100 mmHg), and G3 (Increase to >=100 mmHg). The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments. An increase is defined as an increase in the CTCAE grade relative to the Baseline grade. Participants with missing Baseline values were assumed to have a Baseline value of G0.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  SBP, Increase to Grade 2 | 3
  SBP, Increase to Grade 3 | 0
  DBP, Increase to Grade 2 | 5
  DBP, Increase to Grade 3 | 0

32. Secondary Outcome: Phase II: Number of Participants With Worst-case On-therapy Change From Baseline in Heart Rate
Description: Change from Baseline in heart rate is categorized as decrease to <60 bpm, change to normal or no change, and increase to >100 bpm relative to the Baseline value. Participants with a missing Baseline value are assumed to have a normal Baseline value. Participants were counted twice if the participant's heart rate value decreased to <60 bpm and increased to >100 bpm post-Baseline. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Decrease to <60 bpm | 1
  Change to normal or no change | 4
  Increase to >100 bpm | 1

33. Secondary Outcome: Phase II: Number of Participants With Worst-case On-therapy Change From Baseline in Temperature
Description: Change from Baseline in temperature is categorized as a decrease to <=35 degrees C, change to normal or no change as 35-38 degrees C, and increase to >=38 degrees C relative to the Baseline value. Participants with a missing Baseline value are assumed to have a normal Baseline value. Participants were counted twice if the participant temperature value decreased to <=35 degrees C and increased to >=38 degrees C post-Baseline. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Decrease to <=35 degrees C | 2
  Change to normal or no change | 4
  Increase to >=38 degrees C | 0

34. Secondary Outcome: Phase II: Change From Baseline in Oxygen Saturation Measured Via Pulse Oxymetry at the Indicated Time Points
Description: Oxygen saturation measures the capacity of blood to transport oxygen to other parts of the body. Oxygen binds to hemoglobin in red blood cells when moving through the lungs. A pulse oximeter uses two frequencies of light (red and infrared) to determine the percentage of hemoglobin in the blood that is saturated with oxygen, that is called as blood oxygen saturation, or SpO2. Change from Baseline was calculated as the individual post-Baseline value (Days 8 and 15; Weeks 3 to 132 and post-treatment Visit) minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of oxygen in blood
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Percentage of oxygen in blood
  Day 8, n=6 | -0.2 (0.98)
  Day 15, n=6 | 0.3 (1.51)
  Week 3, n=6 | 0.5 (0.84)
  Week 8, n=6 | 0.5 (1.05)
  Week 12, n=6 | -0.2 (0.98)
  Week 16, n=6 | 0.3 (1.51)
  Week 20, n=5 | -1.0 (1.58)
  Week 24, n=5 | 0.2 (1.64)
  Week 28, n=5 | -0.2 (0.84)
  Week 32, n=5 | -0.6 (1.14)
  Week 36, n=5 | -0.4 (1.34)
  Week 40, n=5 | 0.0 (1.58)
  Week 44, n=4 | -1.3 (2.22)
  Week 48, n=4 | 1.0 (1.41)
  Week 52, n=3 | 1.0 (1.73)
  Week 56, n=3 | -0.7 (0.58)
  Week 60, n=3 | -0.3 (1.15)
  Week 64, n=3 | -0.3 (0.58)
  Week 68, n=3 | 0.0 (1.00)
  Week 72, n=3 | -0.7 (1.53)
  Week 76, n=3 | -1.0 (0.00)
  Week 80, n=3 | 0.0 (1.00)
  Week 84, n=3 | -0.3 (1.53)
  Week 88, n=3 | -0.3 (1.53)
  Week 92, n=3 | 0.3 (0.58)
  Week 96, n=3 | -0.3 (0.58)
  Week 100, n=3 | -0.7 (1.15)
  Week 104, n=3 | -0.3 (1.53)
  Week 108, n=3 | 0.0 (1.00)
  Week 112, n=3 | 0.0 (1.00)
  Week 116, n=3 | -0.7 (0.58)
  Week 120, n=2 | -0.5 (0.71)
  Week 124, n=1 | -2.0 (NA) — There were too few participants to provide a dispersion value.
  Week 128, n=1 | 1.0 (NA) — There were too few participants to provide a dispersion value.
  Week 132, n=1 | -2.0 (NA) — There were too few participants to provide a dispersion value.
  Post-Treatment, n=3 | 1.3 (0.58)

35. Secondary Outcome: Phase II: Change From Baseline in Weight at the Indicated Time Points
Description: Mean change in body weight from baseline was determined. Change from Baseline was calculated as the individual post-Baseline value (Weeks 3 to 132 and post-treatment Visit) minus the Baseline value. The Baseline value is defined as the last pre-treatment value observed.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Kg
  Week 3, n=6 | -0.68 (0.538)
  Week 8, n=6 | -0.22 (0.553)
  Week 12, n=6 | -0.30 (1.273)
  Week 16, n=6 | 0.05 (1.947)
  Week 20, n=5 | -0.32 (2.318)
  Week 24, n=5 | 0.06 (2.243)
  Week 28, n=5 | 0.18 (2.500)
  Week 32, n=5 | 0.42 (2.607)
  Week 36, n=5 | 0.98 (3.016)
  Week 40, n=5 | 0.62 (2.734)
  Week 44, n=4 | 0.80 (3.790)
  Week 48, n=4 | 0.68 (3.527)
  Week 52, n=3 | 1.27 (3.993)
  Week 56, n=3 | 2.23 (3.932)
  Week 60, n=3 | 2.83 (3.879)
  Week 64, n=3 | 2.70 (4.246)
  Week 68, n=3 | 2.87 (4.143)
  Week 72, n=3 | 2.87 (4.165)
  Week 76, n=3 | 3.63 (2.793)
  Week 80, n=3 | 3.43 (4.007)
  Week 84, n=3 | 4.37 (4.008)
  Week 88, n=3 | 3.80 (3.905)
  Week 92, n=3 | 4.13 (3.496)
  Week 96, n=3 | 4.13 (3.630)
  Week 100, n=3 | 3.53 (3.219)
  Week 104, n=3 | 4.00 (4.557)
  Week 108, n=3 | 3.93 (4.800)
  Week 112, n=3 | 3.60 (4.649)
  Week 116, n=3 | 4.20 (4.859)
  Week 120, n=2 | 5.95 (2.192)
  Week 124, n=1 | 7.50 (NA) — There were too few participants to provide a dispersion value.
  Week 128, n=1 | 5.80 (NA) — There were too few participants to provide a dispersion value.
  Week 132, n=1 | 5.30 (NA) — There were too few participants to provide a dispersion value.
  Post-Treatment, n=3 | 0.13 (2.155)

36. Secondary Outcome: Phase II: Number of Participants With the Indicated Electrocardiogram Findings at the Indicated Time Points
Description: Single 12-lead ECGs were performed at Baseline, Weeks 3 to 132 and post-treatment Visit. ECG findings were categorized as: normal, abnormal - CS, or abnormal - NCS, as determined by the investigator.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Baseline, Normal, n=6 | 5
  Baseline, Abnormal-NCS, n=6 | 1
  Baseline, Abnormal-CS, n=6 | 0
  Week 3, Normal, n=6 | 4
  Week 3, Abnormal-NCS, n=6 | 2
  Week 3, Abnormal-CS, n=6 | 0
  Week 12, Normal, n=6 | 4
  Week 12, Abnormal-NCS, n=6 | 2
  Week 12, Abnormal-CS, n=6 | 0
  Week 24, Normal, n=5 | 3
  Week 24, Abnormal-NCS, n=5 | 2
  Week 24, Abnormal-CS, n=5 | 0
  Week 36, Normal, n=5 | 2
  Week 36, Abnormal-NCS, n=5 | 3
  Week 36, Abnormal-CS, n=5 | 0
  Week 48, Normal, n=4 | 3
  Week 48, Abnormal-NCS, n=4 | 1
  Week 48, Abnormal-CS, n=4 | 0
  Week 60, Normal, n=3 | 2
  Week 60, Abnormal-NCS, n=3 | 1
  Week 60, Abnormal-CS, n=3 | 0
  Week 72, Normal, n=3 | 2
  Week 72, Abnormal-NCS, n=3 | 1
  Week 72, Abnormal-CS, n=3 | 0
  Week 84, Normal, n=3 | 1
  Week 84, Abnormal-NCS, n=3 | 2
  Week 84, Abnormal-CS, n=3 | 0
  Week 96, Normal, n=3 | 1
  Week 96, Abnormal-NCS, n=3 | 2
  Week 96, Abnormal-CS, n=3 | 0
  Week 108, Normal, n=3 | 1
  Week 108, Abnormal-NCS, n=3 | 2
  Week 108, Abnormal-CS, n=3 | 0
  Week 120, Normal, n=2 | 1
  Week 120, Abnormal-NCS, n=2 | 1
  Week 120, Abnormal-CS, n=2 | 0
  Week 132, Normal, n=1 | 0
  Week 132, Abnormal-NCS, n=1 | 1
  Week 132, Abnormal-CS, n=1 | 0
  Post-Treatment, Normal, n=3 | 3
  Post-Treatment, Abnormal-NCS, n=3 | 0
  Post-Treatment, Abnormal-CS, n=3 | 0

37. Secondary Outcome: Phase II: Number of Participants With Worst-case On-therapy Change From Baseline in Left Ventricular Ejection Fraction as Assessed by Echocardiogram
Description: Absolute change from Baseline in LVEF were summarized at each scheduled assessment time and in the worst-case post Baseline. Only the post Baseline assessments that used the same method (ECHO or MUGA) as the Baseline assessments were used to derive the change from Baseline. The change from Baseline was categorized as: any increase; no change; 0-<10 Decrease, 10-19 Decrease, >=20 Decrease, >=10 Decrease and >= LLN, >=10 Decrease and below LLN, >=20 Decrease and >=LLN and >=20 Decrease and below LLN. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments.
Time Frame: From Baseline until the post-treatment Visit (average of 1.38 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Number analyzed (Participants) | 6
Participants
  Any Increase | 1
  No change | 0
  0-<10 Decrease | 3
  10-19 Decrease | 2
  >=20 Decrease | 0
  >=10 Decrease and >=LLN | 2
  >=10 Decrease and below LLN | 0
  >=20 Decrease and >=LLN | 0
  >=20 Decrease and below LLN | 0

ADVERSE EVENTS:
Time Frame: On treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of investigational product (IP) until 30 days after the last dose of IP (average of 1.38 years).
Description: SAEs and non-serious AEs were reported for members of the All Treated Subjects (ATS) population, comprised of all participants who had received at least one dose of IP.
Arm/Group | Phase I: GSK2118436 150 mg + GSK1120212 2 mg | Phase II: GSK2118436 150 mg + GSK1120212 2 mg
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: GSK2118436 150 mg + GSK1120212 2 mg (N=6) | Phase II: GSK2118436 150 mg + GSK1120212 2 mg (N=6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: GSK2118436 150 mg + GSK1120212 2 mg (N=6) | Phase II: GSK2118436 150 mg + GSK1120212 2 mg (N=6)
Pyrexia (General disorders) | 5 | 4
Oedema peripheral (General disorders) | 2 | 4
Chills (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 4
Blood alkaline phosphatase increased (Investigations) | 3 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 1 | 1
Blood phosphorus decreased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 2 | 0
Blood albumin decreased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 1 | 0
Glucose urine present (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 2
Bronchitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Paronychia (Skin and subcutaneous tissue disorders) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 3 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Contrast media allergy (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Retinal vascular disorder (Eye disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.